CLINICAL TRIAL: NCT00791648
Title: Short-term Atorvastatin's Effect on Acute Kidney Injury Following Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Frederic T Billings IV, Assistant Professor of Anesthesiology and Critical Care Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 081238
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Acute Kidney Injury; Post-Operative Delirium; Icu Delirium; Acute Renal Failure; Delirium
Keywords: aki; delirium; statin; short-term; cardiac
MeSH Terms: conditions — Acute Kidney Injury; Emergence Delirium; Delirium | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- statin (Experimental): Aim1 intervention: atorvastatin 80mg 1 day prior to open heart surgery and 40mg daily thereafter until hospital discharge.
  Aim2 intervention: atorvastatin 80mg the day of cardiac surgery and 40mg on postop day 1.
  Interventions: Drug: atorvastatin
- placebo (Placebo Comparator): Aim 1 control: placebo one day prior to cardiac surgery and daily thereafter until hospital discharge.
  Aim 2 control: placebo the day of cardiac surgery and postop day 1.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atorvastatin — Aim1 intervention: atorvastatin 80mg 1 day prior to open heart surgery and 40mg daily thereafter until hospital discharge.
  Aim2 intervention: atorvastatin 80mg the day of cardiac surgery and 40mg on postop day 1.
  Other Names: Lipitor
  Arms: statin
Drug: placebo — Aim 1 control: placebo one day prior to cardiac surgery and daily thereafter until hospital discharge.
  Aim 2 control: placebo the day of cardiac surgery and postop day 1.
  Arms: placebo

SUMMARY:
Aim1a: Statin naive patient's scheduled for cardiac surgery will be randomized to 80mg atorvastatin or placebo on the day prior to surgery and then 40mg daily thereafter until hospital discharge to test the hypothesis that short-term atorvastatin use decreases:

1. acute kidney injury following cardiac surgery.
2. postoperative delirium following cardiac surgery.

Aim1b: Patients using statins preoperatively will be randomized to atorvastatin 80mg or placebo on day of surgery and 40mg or placebo on postop day 1 with resumption of preoperative statin therapy on postop day 2 to test the hypothesis that short-term atorvastatin use decreases:

1. acute kidney injury following cardiac surgery.
2. postoperative delirium following cardiac surgery.

Endpoints include glomerular filtration, urine and plasma markers of renal dysfunction, markers of oxidative stress, mitochondrial function, systemic inflammatory markers, delirium, dialysis, stroke, myocardial infarction, time to extubation, ICU length of stay, and death.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery

Exclusion Criteria:

* acute coronary syndrome with troponin leak or unrelenting angina
* liver dysfunction (transaminases 2x normal)
* history of myopathy or liver dysfunction on prior statin therapy
* use of potent CYP3A4 inhibitors such as antifungal azoles, macrolide antibiotics, HIV protease inhibitors, and nefazodone.
* pregnancy or breast feeding
* cyclosporine use
* dialysis
* history of kidney transplant
* fibrate users who cannot stop fibrate use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2009-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic T. Billings, IV, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All study data that are necessary to assess the study hypotheses regarding the primary and secondary outcomes are available for sharing in a manner that protects the privacy of study participants.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available within 6 weeks of request and will be available indefinitely.
Access Criteria: These data will be made available upon reasonable request.

REFERENCES:
- [Derived] Smith LE, Smith DK, Blume JD, Linton MF, Billings FT 4th. High-Density Lipoprotein Cholesterol Concentration and Acute Kidney Injury After Cardiac Surgery. J Am Heart Assoc. 2017 Dec 9;6(12):e006975. doi: 10.1161/JAHA.117.006975. PMID 29223955
- [Derived] Billings FT 4th, Hendricks PA, Schildcrout JS, Shi Y, Petracek MR, Byrne JG, Brown NJ. High-Dose Perioperative Atorvastatin and Acute Kidney Injury Following Cardiac Surgery: A Randomized Clinical Trial. JAMA. 2016 Mar 1;315(9):877-88. doi: 10.1001/jama.2016.0548. PMID 26906014
- [Derived] Billings FT 4th, Ball SK, Roberts LJ 2nd, Pretorius M. Postoperative acute kidney injury is associated with hemoglobinemia and an enhanced oxidative stress response. Free Radic Biol Med. 2011 Jun 1;50(11):1480-7. doi: 10.1016/j.freeradbiomed.2011.02.011. Epub 2011 Feb 18. PMID 21334433

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 patients consented patients were excluded prior to randomization
  14 withdrew, 12 did not require surgery, 4 had unreported baseline live dysfunction, 2 developed acute coronary syndrome, 2 had statin intolerance, 1 died prior to study intervention and surgery, 1 enrolled in another drug study.
Period: Overall Study
Arm/Group | Statin | Placebo
Started | 308 | 309
Completed | 308 | 307
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin | Placebo | Total
Number analyzed (Participants) | 308 | 307 | 615
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [49 to 81] | 67 [51 to 81] | 66 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 94 | 188
  Male | 214 | 213 | 427
Region of Enrollment [Number; unit: participants]
  United States | 308 | 307 | 615

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Kidney Injury
Time Frame: postoperative day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 308 | 307
Participants | 64 | 60
Statistical Analysis 1: Comparison: Statin vs Placebo; Test type: Superiority or Other; p = .75, Pearson x2

2. Primary Outcome: Number of Participants With Delirium
Time Frame: while in ICU (about 2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 308 | 307
Participants | 69 | 75
Statistical Analysis 1: Comparison: Statin vs Placebo; Test type: Superiority or Other; p = .56, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants Requiring Dialysis
Time Frame: while in ICU (about 2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 308 | 307
Participants | 5 | 3
Statistical Analysis 1: Comparison: Statin vs Placebo; Test type: Superiority or Other; p = .71, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Liver Enzyme: Aspartate Aminotransferase Level
Time Frame: postoperative day 1
Measure: Median (95% Confidence Interval); unit: units/liter
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 308 | 307
units/liter | 49 [25 to 105] | 52 [27 to 146]
Statistical Analysis 1: Comparison: Statin vs Placebo; Test type: Superiority or Other; p = .11, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Stroke
Time Frame: while in ICU (about 2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 308 | 307
Participants | 10 | 7
Statistical Analysis 1: Comparison: Statin; Test type: Superiority or Other; p = .06, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants That Died
Time Frame: until postoperative hospital discharge (about 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 308 | 307
Participants | 4 | 1
Statistical Analysis 1: Comparison: Statin vs Placebo; Test type: Superiority or Other; p = .39, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Mitochondrial Function--mtDNA Copy Number
Description: mtDNA copy number
Time Frame: anesthesia induction and POD 1
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: au
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 164 | 168
au
  at anesthesia induction | 0.40 [0.19 to 0.99] | .48 [.21 to 1.1]
  POD 1 | 0.3 [0.17 to 0.3] | 0.43 [0.17 to 0.88]

8. Secondary Outcome: Mitochondrial Function--lactate / Pyruvate Ratio
Description: lactate / pyruvate ratio
Time Frame: anesthesia induction, after CPB, and POD 1
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 80 | 82
ratio
  at anesthesia induction | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.06]
  after CPB | 0.06 [0.03 to 0.09] | 0.06 [0.03 to 0.09]
  POD 1 | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.06]

9. Secondary Outcome: Mitochondrial Function--PGC-1alpha RNA Expression
Description: PGC-1alpha RNA expression
Time Frame: anesthesia induction and POD 1
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: au
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 79 | 76
au
  at anesthesia induction | 0.54 [0.18 to 1.86] | 0.84 [0.23 to 2.51]
  POD 1 | 1.02 [0.27 to 2.45] | 1.37 [0.54 to 3.88]

10. Secondary Outcome: Urine Markers of Renal Injury
Description: tissue inhibitor metaloproteinase-2 x insulin-like growth factor binding protein-7
Time Frame: anesthesia induction, 30 minutes into cardiopulm bypass (CPB), after CPB, ICU admission, 6 hours postop, and Post op Day (POD) 1, 2, 3
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)^2/1000
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 200 | 200
(ng/ml)^2/1000
  at anesthesia induction | 0.119 [0.046 to 0.317] | 0.098 [0.037 to 0.262]
  30 minutes into cardiopulmonary bypass (CPB) | 0.171 [0.062 to 0.442] | 0.169 [0.056 to 0.360]
  after CPB | 0.218 [0.077 to 0.561] | 0.219 [0.087 to 0.619]
  ICU admission | 0.096 [0.043 to 0.238] | 0.112 [0.043 to 0.285]
  6 hours post-op | 0.210 [0.108 to 0.452] | 0.207 [0.084 to 0.438]
  POD 1 | 0.189 [0.040 to 0.489] | 0.186 [0.061 to 0.499]
  POD 2 | 0.170 [0.050 to 0.380] | 0.115 [0.048 to 0.328]
  POD 3 | 0.134 [0.046 to 0.309] | 0.102 [0.054 to 0.287]

11. Secondary Outcome: Plasma Markers of Oxidative Stress: f2-Isoprostanes
Time Frame: anesthesia induction, 30 minutes into cardiopulmonary bypass (CPB), after CPB, ICU admission, 6 hours postop, and POD 1, 2, 3.
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 200 | 200
pg/ml
  at anesthesia induction | 29.4 [20.1 to 41.1] | 28.8 [20.7 to 41]
  30 minutes into cardiopulmonary bypass (CPB) | 41.6 [29.3 to 60.3] | 39 [27.2 to 57.4]
  after CPB | 32.3 [23.6 to 46.8] | 31.5 [23.6 to 45]
  ICU admission | 32.1 [22.1 to 42.4] | 31.6 [23.6 to 44.5]
  6 hours post-op | 32.1 [26.7 to 42.4] | 41 [35.2 to 49]
  POD 1 | 28.1 [21.5 to 39.4] | 30.2 [21.9 to 41.6]
  POD 2 | 28.5 [21.7 to 50.5] | 37 [28 to 47.6]
  POD 3 | 32.7 [27.9 to 54.3] | 26.5 [23.2 to 49.8]

12. Secondary Outcome: Plasma Markers of Oxidative Stress: Isofurans
Time Frame: as for outcome 11
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 200 | 200
pg/ml
  at anesthesia induction | 45 [32.9 to 70] | 48.4 [34.1 to 77.6]
  30 minutes into cardiopulmonary bypass (CPB) | 59.9 [37.9 to 93.8] | 56.2 [42.1 to 89.4]
  after CPB | 57.6 [41.1 to 83.8] | 60.6 [38.1 to 90.2]
  ICU admission | 63.7 [45 to 92.4] | 64 [45.2 to 92.3]
  6 hours post-op | 42.5 [22.5 to 63.9] | 40.4 [29.5 to 59.1]
  POD 1 | 48 [32.1 to 82.5] | 50.9 [34.1 to 85.1]
  POD 2 | 40 [22.8 to 59] | 36 [22 to 46]
  POD 3 | 33.5 [25.3 to 53.9] | 38 [16.5 to 50.2]

13. Secondary Outcome: Urine Markers of Oxidative Stress: f2-Isoprostanes
Time Frame: as for outcome 11
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 178 | 179
ng/mg creatinine
  at anesthesia induction | 1.369 [0.856 to 2.183] | 1.478 [0.836 to 2.237]
  30 minutes into cardiopulmonary bypass (CPB) | 1.750 [0.948 to 2.718] | 2.29 [1.241 to 4.027]
  after CPB | 2.71 [1.247 to 5.38] | 2.729 [1.719 to 4.889]
  ICU admission | 1.816 [0.92 to 03.167] | 2.9 [1.85 to 5.71]
  6 hours post-op | 1.464 [0.839 to 2.389] | 1.77 [1.190 to 3.510]
  POD 1 | 1.056 [0.602 to 1.756] | 1.143 [0.634 to 1.924]
  POD 2 | 0.792 [0.604 to 1.360] | 0.88 [0.7 to 1.548]
  POD 3 | 0.870 [0.527 to 1.601] | 0.875 [0.812 to 1.235]

14. Secondary Outcome: Urine Markers of Oxidative Stress: Isofurans
Time Frame: as for outcome 11
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)^2/1000
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 178 | 178
(ng/ml)^2/1000
  at anesthesia induction | 2.146 [1.321 to 3.316] | 2.146 [1.321 to 3.316]
  30 minutes into cardiopulmonary bypass (CPB) | 2.48 [1.545 to 3.18] | 2.48 [1.545 to 3.18]
  after CPB | 3.709 [2.279 to 6.283] | 3.709 [2.279 to 6.283]
  ICU admission | 3.734 [2.877 to 8.18] | 3.734 [2.877 to 8.18]
  6 hours post-op | 3.310 [1.9 to 5.420] | 3.070 [1.912 to 5.99]
  POD 1 | 2.344 [1.503 to 3.633] | 2.344 [1.503 to 3.633]
  POD 2 | 2.2 [1.428 to 4.050] | 2.2 [1.428 to 4.05]
  POD 3 | 2.16 [1.43 to 2.84] | 2.16 [1.43 to 2.840]

15. Secondary Outcome: Plasma Markers of Inflammation: Measurements of Neuronal Injury (Ubiquitin C-terminal Hydrolase-1)
Description: measurements of neuronal injury (ubiquitin C-terminal hydrolase-1)
Time Frame: anesthesia induction, ICU admission, and POD 1
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 200 | 200
ng/ml
  at anesthesia induction | 6.2 [4.2 to 10] | 6.7 [4.1 to 10.2]
  ICU admission | 12.3 [7.9 to 21.7] | 11.6 [8.0 to 23.9]
  POD 1 | 12.8 [8.3 to 19.5] | 12.2 [8.5 to 17.9]

16. Secondary Outcome: Plasma Markers of Inflammation: Blood Brain Barrier Disruption (S100 Calcium-binding Protein B)
Description: measurements of blood brain barrier disruption (S100 calcium-binding protein B)
Time Frame: anesthesia induction, ICU admission, and POD 1
Population: This marker was only measured in a subset of the total study population, chosen at random.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Statin | Placebo
Number analyzed (Participants) | 200 | 200
pg/ml
  at anesthesia induction | 17.5 [12.5 to 25] | 17 [11.5 to 23.1]
  ICU admission | 163.9 [110.7 to 255.9] | 163.1 [97.3 to 278.5]
  POD 1 | 46.1 [30.4 to 64.2] | 45 [32.7 to 67.9]

ADVERSE EVENTS:
Time Frame: First 10 post-op days
Arm/Group | Statin | Placebo
Serious Adverse Events (participants affected / at risk) | 14/308 | 19/307
Other Adverse Events (participants affected / at risk) | 308/308 | 307/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin (N=308) | Placebo (N=307)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 2 (2)
Severe Infection (Infections and infestations) | 2 (2) | 4 (4)
Severe Peripheral Vascular Ischemia (Vascular disorders) | 1 (1) | 1 (1)
Sternal Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Severe Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hemolytic Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Severe Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Fall with Factured Hip (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Coagulapathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Tamponade (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-operative Injury to Blood Vessel (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Idiopathic Thrombocytopenia Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin (N=308) | Placebo (N=307)
Fever (Infections and infestations) | 50 (125) | 52 (117)
Tachycardia (Cardiac disorders) | 49 (215) | 42 (190)
Hypotension (Cardiac disorders) | 188 (1032) | 192 (1073)
Vasoplegia (Cardiac disorders) | 120 (342) | 118 (357)
Decreased Cardiac Output (Cardiac disorders) | 187 (643) | 194 (623) — Cardiac Output was only measured in patients with a pulmonary artery catheter
Anemia (Surgical and medical procedures) | 183 (1608) | 172 (1537)
Leukocytosis (Infections and infestations) | 141 (513) | 140 (522)
Lactic Acidosis (Cardiac disorders) | 55 (194) | 59 (202)
Transaminemia (Hepatobiliary disorders) | 23 (29) | 39 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes